CLINICAL TRIAL: NCT00870883
Title: Prospective, Randomized, Double-blinded, Placebo-controlled Study of N-acetylcysteine Plus Deferoxamine for Patients With Hypotension as Prophylaxis for Acute Renal Failure
Brief Title: N-acetylcysteine Plus Deferoxamine for Patients With Hypotension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Felipe Dal Pizzol, MD, PhD, Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FR208621
Record Dates: First submitted 2009-03-25; First posted 2009-03-27 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Hypotension; Acute Renal Failure
MeSH Terms: conditions — Hypotension; Acute Kidney Injury | interventions — Acetylcysteine; Deferoxamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- N-acetylcysteine plus deferoxamine (Experimental)
  Interventions: Drug: N-acetylcysteine and deferoxamine

INTERVENTIONS:
Drug: N-acetylcysteine and deferoxamine — N-acetylcysteine bolus dose of 50mg/kg/4h, by a manutention of 100mg/kg/day during 2 days and deferoxamine single dose of 1g administered 15mg/kg/h.

SUMMARY:
Oxidative stress is associated with kidney damage in several different situations, including hypotension. In animal models it has been shown that the combination of n-acetylcysteine plus deferoxamine is superior to its isolate use in the treatment of several diseases. Thus the investigators aimed to determine if the administration of n-acetylcysteine plus deferoxamine could prevent renal failure in critical ill patients who develops hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU
* Presenting hypothesion (MAP < 60mm Hg or the needing to use vasoactive drugs) for at least 30 min in the last 12h before study inclusion

Exclusion Criteria:

* Age lower than 18 years old
* Chronic renal failure
* A known history of allergy to any of the study drugs
* Using n-acetylcysteine to paracetamol overdose
* Pregnant women
* Patients who used iodinated contrast medium
* Hemoglobin less than 6.5 mg/dl
* Cancer patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2009-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Development of acute renal failure | 28 days

SECONDARY OUTCOMES:
28 day-mortality | 28 days
Decrease on plasma oxidative damage and inflammatory parameters | at the end of drug infusion

CONTACTS AND LOCATIONS:
Locations (1):
- São José Hospital, Criciúma, Santa Catarina, Brazil

REFERENCES:
- [Derived] Fraga CM, Tomasi CD, Damasio DC, Vuolo F, Ritter C, Dal-Pizzol F. N-acetylcysteine plus deferoxamine for patients with prolonged hypotension does not decrease acute kidney injury incidence: a double blind, randomized, placebo-controlled trial. Crit Care. 2016 Oct 17;20(1):331. doi: 10.1186/s13054-016-1504-1. PMID 27745551
- [Derived] Fraga CM, Tomasi CD, Biff D, Topanotti MF, Felisberto F, Vuolo F, Petronilho F, Dal-Pizzol F, Ritter C. The effects of N-acetylcysteine and deferoxamine on plasma cytokine and oxidative damage parameters in critically ill patients with prolonged hypotension: a randomized controlled trial. J Clin Pharmacol. 2012 Sep;52(9):1365-72. doi: 10.1177/0091270011418657. Epub 2011 Nov 1. PMID 22045831